CLINICAL TRIAL: NCT01937403
Title: The Use of the Sport Cord Test as a Measure of Physical Performance Following Anterior Cruciate Ligament Reconstruction
Brief Title: Sport Cord Test Following ACL Reconstruction
Status: Completed | Type: Observational
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00003653
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-03

CONDITIONS: Injury of Anterior Cruciate Ligament
Keywords: Physical Therapy; Return to sport
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to determine the interrater reliability and validity of the Sportcord Test as a measure of physical performance following anterior cruciate ligament (ACL) reconstruction. A secondary purpose is to systematically track subjective and objective outcomes on patients following ACL reconstruction to help identify differences between those who have subsequent knee problems and those who do not. The study hypotheses are the following:

1) The Sportcord Test will provide a valid and reliable measure of functional performance following ACL reconstruction. 2) Patients who have subsequent knee problems in the 12 month study period will exhibit different scores on clinical special tests compared to those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgical reconstruction for a torn ACL.
* Returning to participation in a sport(s).
* Will receive physical therapy/rehabilitation after surgical reconstruction for a torn ACL.
* Between ages of 10 and 50.

Exclusion Criteria:

* Non-weight bearing.
* At least 12 weeks removed from surgery.
* Unable to walk, squat, or jump/land without pain in the surgically repaired knee.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients receiving physical therapy/rehabilitation for an ACL surgery and are returning to participation in sports.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2009-10; Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sportcord Test | one year
  The Sportcord Test measures physical performance following an ACL reconstruction. The Sportcord test consists of the following:
  1. single-leg squats
  2. lateral (side-to-side) agility
  3. forward running
  4. backward running

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Shanley, PT, PhD, OCS, CSCS, Principal Investigator — ATI Physical Therapy
Locations (1):
- ATI Physical Therapy, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No